CLINICAL TRIAL: NCT02232399
Title: The Prophylactic Effect of Levosimendan in Reducting Acute Kidney Injury Postoperatively in Pediatric Patients Undergoing Corrective Heart Surgery
Brief Title: Is Levosimendan Superior to Milrinone Regarding Acute Kidney Injury After Cardiac Surgery for Congenital Heart Disease?
Acronym: MiLe-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Albert Castellheim, Associate professor, Göteborg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MiLe-1; 2013-003105-25 (EudraCT Number)
Record Dates: First submitted 2014-09-02; First posted 2014-09-05 (Estimated); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Congenital Heart Defects
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Simendan; Milrinone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Milrinone (Active Comparator): In this arm the patients will receive Milrinone as an inotrope agent. Concentration: 0.2 mg/mL Infusion rate: 0.12 mL / kg / hr = Dose delivered 0.4 μg / kg / min --- Bolus dose: 1.44 ml / kg / hr in ten minutes (a maximum volume 0.24 ml / kg) = 48 μg / kg
  Interventions: Drug: Milrinone
- Levosimendan (Experimental): In this arm the patients will receive Levosimendan as an inotrope agent. Concentration: 0.05 mg/mL Infusion rate: 0.12 mL / kg / hr = Dose delivered 0.1 μg / kg / min --- Bolus dose: 1.44 ml / kg / hr in ten minutes (a maximum volume 0.24 ml / kg) = 12 μg/kg
  Interventions: Drug: Levosimendan

INTERVENTIONS:
Drug: Levosimendan — The drug infusion will be started after initiation of cardiopulmonary bypass and will continue for 24 hours.
  Other Names: Simdax
  Arms: Levosimendan
Drug: Milrinone — The drug infusion will be started after initiation of cardiopulmonary bypass and will continue for 24 hours.
  Other Names: Corotrop
  Arms: Milrinone

SUMMARY:
The aim of the study is to assess the ability of Levosimendan to reduce the postoperative acute kidney injury in pediatric patients undergoing surgery for congenital heart disease (CHDs).

DETAILED DESCRIPTION:
Young children, between the age of 1 to 12 months, with congenital heart disease in need of elective heart surgery will be included in this study.

The trial will contain two study groups, 35 patients in each. One group will receive Levosimendan and the second group will receive Milrinone as a heart muscle-strengthening agent during and after the operation. Milrinone is currently used as the drug of choice in many pediatric cardiac surgery centers. It remains to see if Levosimendan can exert a kidney protecting function in addition to its heart muscle-strengthening properties.

The primary objective of this study is to investigate the preventive effect of Levosimendan on postoperative acute kidney injury in pediatric patients undergoing surgery for their CHDs. Creatinine levels postoperatively will be the primary endpoint. Creatinine, the common marker of kidney injury, will be measured daily.

The treatment with Levosimendan or Milrinone will be started during the operation (after initiation of cardiopulmonary bypass) and will last 24 hours. Blood samples will be obtained at six occasions perioperatively. Patients will be followed 4 days after termination of treatment (totally 5 days).

The duration of study will be 30 days (24 hours treatment + 4 days follow up + 30-days-mortality registration).

Creatinine is the primary outcome in this study. Inflammatory biomarkers and other relevant biomarkers will comprise the secondary outcome variables.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female and male children between 1 and 12 months of age
3. Non-restrictive VSD (corrective surgery)
4. Complete AVSD (biventricular repair)
5. Tetralogy of Fallot

Exclusion Criteria:

1. Unbalanced AtrioVentricular Septal Defect or AVSD with cyanosis
2. Age less than one month and more than one year
3. Acute operation that is unscheduled operation during the first 24 hours after presentation to the department for thoracic surgery
4. Mild, moderate, or severe kidney dysfunction and known anatomical anomalies of kidneys
5. Liver impairment or disease
6. Ongoing infection
7. Use of nephrotoxic drugs (like ibuprofen, angiotensin-converting-enzyme inhibitors, gentamicin, vancomycin) preoperative or postoperative until first post operative day. Contrast agents whithin 24 hours before operation.
8. Use of inhibitors of membrane transport proteins (cimetidine, cetirizine, trimethoprim, probenecid, rifampin and gemfibrosil).
9. Allergy to Levosimendan or substance included in the preparation or previous use of Levosimendan.
10. Severe arrhythmias needing pace-maker treatment prior to the operation
11. Severe cardiac dysfunction needing for treatment with extracorporeal membrane oxygenation (ECMO) prior to the operation.
12. Preoperative need for mechanical ventilation and/or inotropic agents.
13. Re-operation (open heart surgery). Earlier surgical closure of the arterial duct does not count as an exclusion criteria.
14. Prematurity: Gestational age < 30 weeks, irrespective of postpartum age. Gestational age 30-34 weeks if patient is included at postpartum age under 3 months.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Castellheim, MD, PhD, Principal Investigator — Queen Silvia Children´s Hospital, Department of anesthesia and intensive care; Håkan Wåhlander, MD, PhD, Study Chair — Queen Silvia Children´s Hospital, Department of pediatric cardiology; Birgitta Romlin, MD, PhD, Study Chair — Queen Silvia Children´s Hospital, Department of anesthesiology and intensive care; Elin Thorlacius, MD, Study Chair — Queen Silvia Children´s Hospital, Department of anesthesiology and intensive care; Sven-Erik Ricksten, MD, PhD, Study Chair — Sahlgrenska University Hospital, Department of anesthesiology and intensive care
Locations (2):
- Children´s Hospital, Helsinki University Central Hospital, Helsinki, Finland
- Queen Silvia Children´s Hospital, Gothenburg, Västra Götaland County, Sweden

REFERENCES:
- [Derived] Thorlacius EM, Vistnes M, Ojala T, Keski-Nisula J, Molin M, Romlin BS, Synnergren M, Ricksten SE, Wahlander H, Castellheim A. Levosimendan Versus Milrinone and Release of Myocardial Biomarkers After Pediatric Cardiac Surgery: Post Hoc Analysis of Clinical Trial Data. Pediatr Crit Care Med. 2021 Jul 1;22(7):e402-e409. doi: 10.1097/PCC.0000000000002712. PMID 33739957

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Assessed for eligibility (n= 123)
  Excluded (n=51)
  * Lack of informed consent (n=15)
  * Other exclusion criteria (n=21)
  * Study personnel not available (n=14)
  * Patient moved to another center (n=1)
  Randomized (n= 72)
Groups:
- Milrinone: Allocated to milrinone (n=39)
  • Received allocated intervention (n=39) Did not receive allocated intervention (n=0)
- Levosimendan: Allocated to levosimendan (n=33)
  * Received allocated intervention (n=32)
  * Did not receive allocated intervention (n=1, consent withdrawn)
Period: Overall Study
Arm/Group | Milrinone | Levosimendan
Started | 39 | 33
Completed | 38 | 32
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Milrinone | Levosimendan | Total
Number analyzed (Participants) | 38 | 32 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 38 | 32 | 70
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: Months] | 5.6 (2.7) | 5.9 (2.9) | 5.6 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 36
  Male | 18 | 16 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 14 | 18 | 32
  Finland | 24 | 14 | 38
S-Creatinine [Mean (Standard Deviation); unit: μmole/L] | 23.9 (6.1) | 25.9 (5.9) | 24.5 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: S-creatinine
Description: The primary outcome variable was the absolute value of serum creatinine data on postoperative day 1.
Time Frame: One day after cardiac surgery
Measure: Mean (Standard Deviation); unit: μmol/L
Groups:
- Milrinone: Patients who received milrionen
- Levosimendan: Patients who received levosimendan
Arm/Group | Milrinone | Levosimendan
Number analyzed (Participants) | 38 | 32
μmol/L
  Preoperative | 23.9 (6.1) | 25.9 (5.9)
  Postop day 1 | 33.7 (12.9) | 34.2 (2.0)
Statistical Analysis 1: Comparison: Milrinone vs Levosimendan; To test whether there were any significant differences between the two treatment groups over time (group vs time interaction), a repeated measurement mixed-model approach was used. This assumed an unstructured covariance pattern; Test type: Other; p = 0.45, Mixed Models Analysis — To test whether there were any significant differences between the two treatment groups over time (group vs time interaction), a repeated measurement mixed-model approach was used. This assumed an unstructured covariance pattern; Unstructured covariance pattern was assumed

2. Secondary Outcome: Acute Kidney Injury (AKI)
Description: Secondary outcomes included the occurrence rate of AKI, defined as a 50% rise in serum creatinine, or more, within 48 hours after surgery. All stages of AKI (stage 1 and stage 2 and stage 3)
Time Frame: Two days (second postoperative day)
Measure: Count of Participants; unit: Participants
Groups:
- Milrinone: Patients who received milrinone
Arm/Group | Milrinone | Levosimendan
Number analyzed (Participants) | 38 | 32
Participants | 15 | 15
Statistical Analysis 1: Comparison: Milrinone vs Levosimendan; Test type: Other; p = 0.70, Regression, Logistic

3. Secondary Outcome: 30 Days Mortality
Description: Mortality at 30th day
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Milrinone | Levosimendan
Number analyzed (Participants) | 38 | 32
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days
Arm/Group | Milrinone | Levosimendan
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/32
Serious Adverse Events (participants affected / at risk) | 6/38 | 9/32
Other Adverse Events (participants affected / at risk) | 11/38 | 8/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milrinone (N=38) | Levosimendan (N=32)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) — Nodal tachycardia and low cardiac output syndrome postoperatively. Re-operation on the first operative night; Study drug was stopped on the first postoperative night and the patient was excluded from the study
Pericardial fluid and sepsis (Cardiac disorders) | 1 (1) | 0 (0) — Prolonged hospital stay due to: 1) Operation for pericardial fluid drainage 2) treatment for sepsis with antibiotics
Pericard effusion (Cardiac disorders) | 1 (1) | 0 (0) — Prolonged hospital stay due to: Pericardiac drainage on postop day 11, due to pericardial effusion
Verified bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) — Prolongation of existing hospitalization due to verified bacterial sepsis (Staphylococcus aureus)
Closure of another small VSD + tricuspid valve plasty + permanent pacemaker due to total AV-block (Cardiac disorders) | 1 (1) | 0 (0) — Prolonged hospital stay due to two re-operations; first for closure of another small VSD and tricuspid valve plastic, and second for inserting permanent pacemaker due to total AV-block.
Readmission for pericardal fluid drainage (Cardiac disorders) | 1 (1) | 0 (0) — Readmission due to pericardial fluid and re-operation for drainage of the fluid.
Readmission (Cardiac disorders) | 0 (0) | 1 (1) — Readmission on postop day 20 due to common cold and vomiting.
Re-operation and dialysis post re-operation (Cardiac disorders) | 0 (0) | 1 (1) — Prolonged hospitalisation due to re-operation on postop day 6 and prolonged PICU stay after re-operation. Peritoneal dialysis for total 11 days.
Enalapril caused prolonged hospitalisation (Cardiac disorders) | 0 (0) | 1 (1) — Increased creatinine and increased need for diuretics. Patient recovered when enalapril was removed.
Fever and diarrea (Infections and infestations) | 0 (0) | 1 (1) — Fever and diarrhoea in ward on postoperative day 8. High CRP but negative blood cultures. Was treated as sepsis.
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) — Prolonged hospital stay due to Upper respiratory infection postoperatively in PICU
AV block III (Cardiac disorders) | 0 (0) | 1 (1) — AV block III, received permanent pacemaker
Blood culture verified S. aureus sepsis (Infections and infestations) | 0 (0) | 1 (1) — Prolonged hospitalisation due to blood culture verified S. aureus sepsis.
Postoperative AV-block (Cardiac disorders) | 0 (0) | 1 (1) — AV-block Episodes postoperatively, received permanent pace-maker 4 months after the operation
hydrocephalus and seizure (Nervous system disorders) | 0 (0) | 1 (1) — hydrocephalus and bleeding from an old cerebral infarction. Ventriculostomy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Milrinone (N=38) | Levosimendan (N=32)
Inotropic score > 20 (Nervous system disorders) | 4 | 3
Junctional ectopic tachycardia (Cardiac disorders) | 7 | 3
Third-degree atrioventricular block (Cardiac disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
1. The trial included merely three types of heart defects with relatively short CPB-times.

   Patient with higher risk for postoperative AKI were excluded (patients with univentricular circulation, renal disease, history of open-heart surgery or receiving nephrotoxic agents
2. Unequal number of patients in the study groups (due to use of the stratification program which was set to stratify the patients according to age and diagnosis).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT02232399/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT02232399/SAP_001.pdf